CLINICAL TRIAL: NCT06890117
Title: Non-surgical Treatment of Peri-implantitis Using Combined Er: YAG (2940nm) and Diode Laser (808nm): a Randomized Controlled Clinical Trial. Clinical, Microbiological Parameters and Metabolomics
Brief Title: Non-Surgical Laser Treatment for Peri-Implantitis: Er:YAG & Diode Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26/29.01.2025
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Peri-Implantitis
Keywords: Non-surgical therapy; Er:YAG laser; Diode laser; Microbiological analysis; Metabolomics; RCT
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a control group receiving non-surgical ultrasonic debridement and an experimental group receiving Er:YAG and Diode laser treatment.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor evaluating clinical and microbiological parameters will be blinded to the treatment allocation to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic Debridement + Saline Irrigation (Active Comparator): Participants in this group will receive non-surgical mechanical debridement using ultrasonic scalers specifically designed for implant surfaces, followed by irrigation with saline solution. No additional laser therapy will be applied.
  Interventions: Device: Ultrasonic Scalers with EMS PI tip and Saline Irrigation
- Er:YAG + Diode Laser (Experimental): Participants in this group will receive non-surgical peri-implantitis treatment using Er:YAG (2940 nm) and Diode (808 nm) lasers. The Er:YAG laser will be used for implant surface decontamination, while the Diode laser will be applied for biostimulation.
  Interventions: Device: Er:YAG (2940nm) and Diode (808nm) Laser

INTERVENTIONS:
Device: Ultrasonic Scalers with EMS PI tip and Saline Irrigation — Control Group: Non-surgical peri-implantitis treatment using ultrasonic scalers and EMS PI tips designed for implants, combined with saline irrigation to remove plaque and biofilm from implant surfaces.
  Other Names: Ultrasonic Debridement
  Arms: Ultrasonic Debridement + Saline Irrigation
Device: Er:YAG (2940nm) and Diode (808nm) Laser — Experimental Group: Non-surgical peri-implantitis treatment using Er:YAG laser (2940nm) and Diode laser (808nm) for decontamination of the implant surface and surrounding tissues. The Er:YAG laser is used for mechanical debridement and biofilm removal, while the Diode laser has biostimulatory effects.
  Other Names: Laser-Assisted Peri-Implantitis Treatment
  Arms: Er:YAG + Diode Laser

SUMMARY:
A prospective, randomized clinical trial with a 3-month duration was designed to evaluate the efficacy of non-surgical treatment for peri-implantitis. Patients presenting at the Postgraduate Periodontology Clinic of the School of Dentistry, Aristotle University of Thessaloniki, with a diagnosis of peri-implantitis in at least one implant (based on the new classification of periodontal and peri-implant diseases, EFP 2018) will be included.

After clinical and radiographic evaluation, patients will be randomly assigned to two groups, with each patient participating in the study with one implant. The control group will receive non-surgical treatment using ultrasonic scalers designed for implants, combined with saline irrigation. The experimental group will undergo non-surgical treatment with Er:YAG (2940nm) and Diode (808nm) laser. All patients will receive oral hygiene instructions at baseline and during each subsequent visit.

Microbial plaque samples will be collected using two sterile paper cones from the deepest peri-implant pocket before treatment and three months after treatment. The presence and absolute counts of Porphyromonas gingivalis and Filifactor alocis will be assessed using quantitative polymerase chain reaction (qPCR). Additionally, peri-implant crevicular fluid will be collected from the second deepest peri-implant pocket using three sterile paper cones before treatment and three months post-treatment for metabolomic analysis.

Clinical parameters, including probing pocket depth (PPD), bleeding on probing (BOP), clinical attachment level (CAL), peri-implant mucosal recession (REC), and suppuration (SUP), will be recorded at baseline and at the end of the experimental period (3 months). Treatment success will be evaluated at the 3-month mark, defined as a pocket depth ≤5 mm with no bleeding on probing at more than one of six implant sites and no suppuration, according to the EFP S3 level clinical practice guideline.

Additionally, patients will complete a home questionnaire to assess pain at different time points (immediately after treatment, 24, 48, and 72 hours post-treatment). Pain levels will be evaluated using a 100-mm visual analog scale (VAS), where 0 mm indicates "no pain" and 100 mm represents "worst pain." The total number of analgesics consumed daily for one week post-treatment will also be recorded. At the end of the week, patients will answer four Yes/No/Don't Know questions to assess their satisfaction with the treatment.

DETAILED DESCRIPTION:
This study aims to compare the effectiveness of non-surgical peri-implantitis treatment using conventional ultrasonic debridement versus a laser-assisted approach. The primary objective is to assess clinical, microbiological, and metabolomic outcomes associated with each treatment modality.

The study will be conducted at the Postgraduate Periodontology Clinic of the School of Dentistry, Aristotle University of Thessaloniki. Participants will be screened based on inclusion and exclusion criteria, and those diagnosed with peri-implantitis in at least one implant will be randomly assigned to either the control or experimental group.

Study Procedures:

Control Group: Treatment with ultrasonic scalers designed for implants and saline irrigation.

Experimental Group: Treatment with Er:YAG (2940nm) and Diode (808nm) laser.

Oral Hygiene Instructions: Provided at baseline and each follow-up visit.

Microbiological Sampling: Collection of subgingival plaque using sterile paper cones before and after treatment (3 months), with analysis of P. gingivalis and F. alocis using qPCR.

Metabolomic Analysis: Collection of peri-implant crevicular fluid before and after treatment for metabolomic profiling.

Clinical Parameters: PPD, BOP, CAL, REC, and SUP will be recorded at baseline and after 3 months.

Pain and Patient Satisfaction: VAS pain assessment at multiple time points and tracking of analgesic consumption. A patient satisfaction questionnaire will be completed at the end of the study.

Study Outcomes:

Primary Outcome: Reduction in peri-implant pocket depth and inflammation.

Secondary Outcomes: Changes in microbiological and metabolomic markers, pain perception, and patient-reported satisfaction.

This randomized controlled clinical trial aims to provide valuable insights into the efficacy of laser-assisted non-surgical therapy for peri-implantitis compared to conventional ultrasonic debridement. The findings could contribute to the optimization of non-surgical treatment protocols for peri-implant disease management.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the Postgraduate Periodontology Clinic with a diagnosis of peri-implantitis in at least one implant, based on the 2018 Classification of Periodontal and Peri-Implant Diseases (EFP 2018).
* Probing pocket depth (PPD) of up to 10 mm.
* Periodontally healthy individuals (no active periodontal disease).
* Implants must have been in function (loaded) for at least one year.
* Age ≥ 18 years.
* Medically healthy individuals or those with well-controlled systemic conditions.
* Implant-supported restorations must be accessible for proper oral hygiene.
* Patients must provide signed informed consent for participation.
* Non-smokers only

Exclusion Criteria:

* Presence of systemic diseases or medications that could influence treatment outcomes (e.g., uncontrolled diabetes, chemotherapy, immunosuppression).
* Underwent peri-implantitis treatment in the past 3 months.
* Use of antibiotics or antimicrobial therapy in the past 3 months.
* Pregnancy or breastfeeding.
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) | Baseline and 3 months post-treatment
  Change in peri-implant probing pocket depth (PPD) from baseline to 3 months post-treatment. PPD is measured using a periodontal probe at six sites per implant.

SECONDARY OUTCOMES:
Bleeding on Probing (BOP) | Baseline and 3 months post-treatment
  Assessment of bleeding upon gentle probing at six sites per implant to evaluate inflammation.
Clinical Attachment Level (CAL) | Baseline and 3 months post-treatment
  Measurement of the distance from the implant shoulder to the base of the peri-implant pocket.
Peri-implant Mucosal Recession (REC) | Baseline and 3 months post-treatment
  Measurement of the vertical soft tissue recession at six implant sites.
Presence of Suppuration (SUP) | Baseline and 3 months post-treatment
  Assessment of purulent exudate upon probing, indicating ongoing infection.
Treatment Success (Yes/No) | 3 months post-treatment
  Defined as pocket depth ≤5 mm with no bleeding on probing at more than one of six implant sites and no suppuration, per EFP S3 guidelines.
Change in P. gingivalis Levels | Baseline and 3 months post-treatment
  Quantification of Porphyromonas gingivalis using qPCR from subgingival plaque samples.
Change in F. alocis Levels | Baseline and 3 months post-treatment
  Quantification of Filifactor alocis using qPCR from subgingival plaque samples.
Metabolomic Profile Changes | Baseline and 3 months post-treatment
  Analysis of peri-implant crevicular fluid metabolites to assess biochemical changes post-treatment.
Pain Evaluation (VAS Scale) | 0, 24, 48, and 72 hours post-treatment
  Pain assessment using a 100-mm Visual Analog Scale (VAS) at different time points (immediately post-treatment, 24, 48, and 72 hours). The VAS for Pain ranges from 0 to 100, where 0 represents no pain and 100 represents the worst possible pain. Higher scores indicate greater pain severity.
Analgesic Consumption | Daily for 7 days post-treatment
  Total number of analgesics taken by patients in the first week post-treatment.
Patient Satisfaction | 1 week post-treatment
  Yes/No/Don't Know questionnaire assessing patient satisfaction with treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia Neofytou, MSc, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study, including clinical data (e.g., probing pocket depth, bleeding on probing), microbiological data (e.g., counts of P. gingivalis and F. alocis), and metabolomics data, will be made available to other researchers after the study's completion. This data will be shared for the purpose of further analysis, with a focus on advancing research in peri-implantitis and dental treatments.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The individual participant data, along with the supporting information, will become available after the publication of the final results of this study. The exact timeline for availability and duration of access has not yet been decided.
Access Criteria: The access criteria for the individual participant data (IPD) and supporting information have not yet been decided. Further details regarding the review process, who will have access, and the types of analyses permitted will be determined after the publication of the final study results.

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Camps-Font O, Perez-Beltran I, Fornes-Nieto V, Gonzalez-Barnadas A, Costa-Berenguer X, Garcia-Garcia M, Figueiredo R, Valmaseda-Castellon E. Patient-centered outcomes after surgical treatment of peri-implantitis: a prospective clinical study. Med Oral Patol Oral Cir Bucal. 2023 Jan 1;28(1):e72-e80. doi: 10.4317/medoral.25587. PMID 36243998
- [Background] Grzech-Lesniak K, Sculean A, Gaspirc B. Laser reduction of specific microorganisms in the periodontal pocket using Er:YAG and Nd:YAG lasers: a randomized controlled clinical study. Lasers Med Sci. 2018 Sep;33(7):1461-1470. doi: 10.1007/s10103-018-2491-z. Epub 2018 May 15. PMID 29766330
- [Background] Mills MP, Rosen PS, Chambrone L, Greenwell H, Kao RT, Klokkevold PR, McAllister BS, Reynolds MA, Romanos GE, Wang HL. American Academy of Periodontology best evidence consensus statement on the efficacy of laser therapy used alone or as an adjunct to non-surgical and surgical treatment of periodontitis and peri-implant diseases. J Periodontol. 2018 Jul;89(7):737-742. doi: 10.1002/JPER.17-0356. No abstract available. PMID 29693260
- [Background] Schwarz F, Aoki A, Becker J, Sculean A. Laser application in non-surgical periodontal therapy: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):29-44. doi: 10.1111/j.1600-051X.2008.01259.x. PMID 18724840
- [Background] Schwarz F, Sculean A, Georg T, Reich E. Periodontal treatment with an Er: YAG laser compared to scaling and root planing. A controlled clinical study. J Periodontol. 2001 Mar;72(3):361-7. doi: 10.1902/jop.2001.72.3.361. PMID 11327064
- [Background] Schwarz F, Sculean A, Rothamel D, Schwenzer K, Georg T, Becker J. Clinical evaluation of an Er:YAG laser for nonsurgical treatment of peri-implantitis: a pilot study. Clin Oral Implants Res. 2005 Feb;16(1):44-52. doi: 10.1111/j.1600-0501.2004.01051.x. PMID 15642030